CLINICAL TRIAL: NCT03818061
Title: A European, Multi-centre Phase II Trial of Atezolizumab and Bevacizumab in Patients With Recurrent or Metastatic Squamous-cell Carcinoma of the Head and Neck (HNSCC)
Brief Title: Atezolizumab and Bevacizumab in Patients With Recurrent or Metastatic Squamous-cell Carcinoma of the Head and Neck
Acronym: ATHENA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET 18-156 ATHENA
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Neoplasms
Keywords: Atezolizumab; Bevacizumab
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: The sample size calculation will use an adaptive Simon 2-stage design based on the strategy developed by Lin and Shih (Biometrics 2004). This method allows checking the result at the first stage, adjusting the power and success rate if necessary, and adapting the decision rule accordingly. A minimum of 69 patients (up to 110) will be enrolled in 2 parallel independent cohorts depending on the HPV status of their tumors: cohort A (HPV+, N = 42 to 59) and cohort B (HPV-, N = 27 to 51).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV + (Experimental): Patient with Human papillomavirus (HPV +) treated by Atezolizumab combined with Bevacizumab.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- HPV - (Experimental): Patient without Human papillomavirus (HPV - ) treated by Atezolizumab combined with Bevacizumab.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Patients will receive the combination of Atezolizumab 1200 mg and Bevacizumab 15 mg/kg by IV infusion every 3 weeks.
  Other Names: Tecentriq
Drug: Bevacizumab — Patients will receive the combination of Atezolizumab 1200 mg and Bevacizumab 15 mg/kg by IV infusion every 3 weeks.
  Other Names: Avastin

SUMMARY:
This proof-of-concept study aims to assess the clinical and biological effects of Atezolizumab combined with Bevacizumab in advanced previously treated squamous-cell carcinoma of the head and neck (HNSCC).

DETAILED DESCRIPTION:
Patients will receive the combination of Atezolizumab 1200 mg and Bevacizumab 15 mg/kg by IV infusion every 3 weeks. Treatment will be continued until disease progression, unacceptable toxicity or voluntary withdrawal. In the absence of unacceptable toxicity, patients who meet criteria for disease progression per RECIST v1.1 while receiving study treatment will be permitted to continue the study treatment if they meet all of the following criteria:

* Evidence of clinical benefit, as determined by the investigator following a review of all available data
* Absence of symptoms and signs (including laboratory values, such as new or worsening hypercalcemia) indicating unequivocal progression of disease
* Absence of decline in ECOG Performance Status that can be attributed to disease progression
* Absence of tumor progression at critical anatomical sites (e.g., leptomeningeal disease) that cannot be managed by protocol-allowed medical interventions.

ELIGIBILITY:
Inclusion Criteria:

I1. Male or female patient ≥18 years of age at time of informed consent form signature.

I2. Histologically proven advanced/metastatic HNSCC (oropharynx, oral cavity, hypopharynx and larynx). Patients with cancer of nasopharynx (i.e. cavum cancer) are not eligible.

I3. Documented radiological progression or relapse after platinum-containing systemic therapy in the advanced/metastatic setting. Patients may have received anti-EGFR agents (in combination or sequential) and other standard first-line treatment for metastatic HNSCC available at time of enrolment.

I4. Documented tumor HPV status (positive and negative are eligible) based on p16 IHC testing by local testing.

I5. Measurable disease at baseline according to RECIST V1.1. Note: Lesions intended to be biopsied should not be defined as target lesions. I6. Availability of a representative formalin-fixed paraffin-embedded (FFPE) primary and/or metastatic tumor tissue with an associated pathology report from an archival block.

I7. Optional : Tumor lesion visible by medical imaging and accessible to repeatable percutaneous or endoscopic sampling that permits core needle biopsy without unacceptable risk of a significant procedural complications, and suitable for retrieval of 4 cores with a needle minimum diameter :16-gauge.

I8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1. I9. Life expectancy > 18 weeks.

I10. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 7 days prior to C1D1:

* Bone marrow (without transfusion within 2 weeks before C1D1)

  * WBC ≥ 2.5 x 109/L
  * Hemoglobin ≥ 9.0 g/dL. Patients may be transfused (> 2 weeks before C1D1) to meet this criterion.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without granulocyte colony-stimulating factor support within 2 weeks before C1D1.
  * Platelets ≥ 100 x 109/L
  * Lymphocyte count ≥ 0.5 x 109/L
* Renal function

  -Serum creatinine clearance ≥30 mL/min/1.73m2 (MDRD or CKD-EPI formula) or serum creatinine ≤1.5ULN.
* Hepatic function

  * Serum bilirubin ≤ 1.5 × Upper Limit of Normal (ULN), with the following exception: Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 2.5 x ULN, with the exceptions of patients with liver involvement for whom AST and/or ALT and/or PAL ≤ 5 ULN is acceptable.
* Coagulation

  * Prothrombin time/INR ≤ 1.5, or, if patient is receiving therapeutic anticoagulation, prothrombin time/INR < 3.0
  * aPTT ≤ ULN OR, if patient is receiving therapeutic anticoagulation, aPTT must be < 1.5 ULN.
* Proteinuria by urine dipstick < 2+ or 24-hour proteinuria ≤ 1.0 g. I11. Women patients of child-bearing potential are eligible, provided they have a negative serum or urine pregnancy test within 7 days prior to C1D1, and agrees to use adequate contraception (for example, intrauterine device [IUD], birth control pills unless clinically contraindicated, or barrier device) beginning 2 weeks before the first dose of study drugs and for up to 6 months after the final dose of study drugs.

I12. Fertile men must agree to use an effective method of contraception during the study and for up to 6 months after the last dose of study drugs.

I13. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed and should be able and willing to comply with study visits and procedures as per protocol.

I14. Patients must be covered by a medical insurance in country where applicable.

Exclusion Criteria:

E1. Malignancies other than HNSCC within 3 years prior to C1D1 with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localised prostate cancer or ductal carcinoma in situ treated surgically with curative intent).

E2. More than two prior lines of systemic therapy for recurrent or metastatic HNSCC.

E3. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

Note: Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:

* Measurable disease, per RECIST v1.1, must be present outside the CNS.
* The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
* Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
* There is no evidence of interim progression between completion of CNS-directed therapy and initiation of study treatment.
* The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, neurosurgical resection within 28 days prior to initiation of study treatment.
* The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted.
* Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.

E4. Evidence of tumor lesion is hemorrhagic or radiographic evidence of major blood vessel invasion/infiltration of tumor demonstrating >90° abutment or encasement of a major blood vessel.

E5. Spinal cord compression not definitively treated with surgery and/or radiation.

E6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.

E7. Uncontrolled tumor pain.

* Patients who require narcotic pain medication during screening should be on a stable dose regimen prior to C1D1.
* Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to C1D1. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
* Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.

E8. Acute and ongoing toxicities from previous therapy that have not resolved to Grade ≤ 1, except for alopecia, neuropathy and lab values presented in inclusion criteria.

E9. Prior treatment with CD137 agonists or immune checkpoint blockade therapies (including PD-1 and PD-L1, CTLA4 inhibitors), or with VEGF/VEGFR inhibitors.

E10. Prior allogeneic bone marrow transplantation or solid organ transplant for another malignancy in the past.

E11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to C1D1, or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to C1D1 or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure.

E12. Prior radiation therapy within 21 days prior to C1D1 and/or persistence of radiation-related Grade > 1 AE (including CNS radiotherapy and palliative radiotherapy according to E3 and E8).

E13. Treatment with any investigational agent or approved anti-cancer therapy within 28 days or five investigational agent half-lives (whichever is longer) prior to C1D1.

E14. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to C1D1, or anticipation of need for systemic immunosuppressive medication during study treatment; with the exceptions of intranasal,inhaled or topical corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.

E15. Systemic immunostimulatory agents (including, but not limited to, interferons and IL-2) are prohibited within 4 weeks or five half-lives of the drug (whichever is longer) prior to C1D1.

E16. Oral or IV antibiotics within 14 days of C1D1. Note: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible.

E17. Use within 10 days prior to C1D1 of the following treatment:

* Acetylsalicylic acid (> 325 mg/day) (Note: lower dose is acceptable before and during the treatment period).
* Clopidogrel (> 75 mg/day) (Note: lower dose is acceptable before and during the treatment period)
* Therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes except if INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks at C1D1.

E18. History of severe allergic or other hypersensitivity reactions to:

* chimeric or humanized antibodies or fusion proteins,
* biopharmaceuticals produced in Chinese hamster ovary cells, or
* any component of the Atezolizumab or Bevacizumab formulations E19. Concurrent treatment with any other anti-cancer treatment, approved or investigational agent or participation in another clinical trial with therapeutic intent.

E20. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis with the following exceptions:

* patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone,
* patients with controlled Type 1 diabetes mellitus,
* patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * rash must cover less than 10% of body surface area (BSA).
  * disease is well controlled at baseline and only requiring low potency topical steroids.
  * no acute exacerbations of underlying condition within the previous 12 months requiring PUVA (Psoralen plus Ultraviolet A radiation), methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high-potency or oral steroids"

E21. Infectious diseases :

* active infection requiring IV antibiotics,
* severe infection within 4 weeks prior to C1D1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia,
* active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening), Note : Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to C1D1.
* active hepatitis C. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA at screening
* HIV infection,
* active tuberculosis
* influenza vaccination should be given during influenza season. Patients must not receive live attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to C1D1 or at any time during the study.

E22. Significant cardiovascular disease :

* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to C1D1, unstable arrhythmias, acute coronary syndromes (including unstable angina), or history of coronary angioplasty/stenting/bypass grafting within past 6 months.
* Left Ventricular Ejection Fraction (LVEF) < 40% at screening.
* Known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Severe cardiac arrhythmia requiring medication or severe conduction abnormalities
* Clinically significant valvular disease, cardiomegaly, ventricular hypertrophy, or cardiomyopathy.
* Uncontrolled hypertension defined by systolic pressure > 150 mm Hg and/or diastolic pressure > 100 mm Hg, with or without anti-hypertensive medication. Patients with initial blood pressure elevations are eligible if initiation or adjustment of anti-hypertensive medication lowers blood pressure to meet entry criteria.
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of stroke or transient ischemic attack within 6 months prior to C1D1
* Clinically significant peripheral vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to C1D1.

E23. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.

E24. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to C1D1.

E25. Serious non-healing wound, active ulcer or untreated bone fracture. E26. History of hemoptysis (≥ ½ teaspoon of bright red blood per episode), or any other serious hemorrhage or at risk of bleeding (gastrointestinal history of bleeds, gastrointestinal ulcers, etc.).

E27. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding.

E28. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).

E29. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At 18 weeks
  Overall response rate (ORR), defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR), on two consecutive occasions at least 4 weeks apart, determined by investigator per RECIST v1.

SECONDARY OUTCOMES:
Disease control rate | At 18 weeks
  Disease control rate (DCR) defined as the proportion of patients with Complete Response (CR), Partial Response (PR) or Stable Disease (SD) at 18 weeks determined by investigator per RECIST v1.1
Best Overall Response Rate | Every 6 weeks for 2 years then every 9 weeks for 3 years
  Best Overall Response Rate (BORR) is determined by the best response designation recorded between the date of the first study treatment and the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first.
Duration of response | Every 6 weeks for 2 years then every 9 weeks for 3 years
  Duration of response (DoR), defined as the time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression or death is documented, whichever occurs first.
Progression-free survival | Every 6 weeks for 2 years then every 9 weeks for 3 years
  Progression-free survival (PFS), defined as the time from the first day of study treatment to the date of the first documented tumor progression or death due to any cause, whichever occurs first.
Overall survival | Up to 1 year
  Overall survival (OS) is the time from the first day of study treatment to the date of death due to any cause.
HPV+ vs HPV - | At Baseline, at cycle 3 (each cycle is 21 days) and in case of relapse for 2 years
  Exploratory analyses on tumor biopsy samples include molecular characterization and comparison of HPV+ versus HPV- tumors and tumor microenvironment.
PD1-/PD-L1 expression | At Baseline, at cycle 3 (each cycle is 21 days) and in case of relapse for 2 years
  Exploratory analyses on tumor biopsy samples include PD1-/PD-L1 expression at baseline and after treatment by IHC/IF on tumor cells and immune infiltrate and correlation to soluble forms determined by ELISA in blood samples.
Immune cells infiltrate characterization | At Baseline, at cycle 3 (each cycle is 21 days) and in case of relapse for 2 years
  Exploratory analyses on tumor biopsy samples include Immune cells infiltrate characterization.
Immuno-phenotyping | At Baseline, at Cycle 1 day 7 (each cycle is 21 days), cycle 2, cycle 3 and in case of relapse for 2 years
  Exploratory analyses on blood samples include immuno-phenotyping.
Cytokines Production | At Baseline, at Cycle 1 day 7 (each cycle is 21 days), cycle 2, cycle 3 and in case of relapse for 2 years
  Exploratory analyses on blood samples include cytokines production by blood T cells (using DMSO cryopreserved PBMCs) according to ICP receptor expression. Intracytoplasmic cytokines will be measured after PMA/ionomycin restimulation by multi-parametric flow cytometry. The response will be determined according PD-1 versus other ICP expression.
Microbiome analysis | At Baseline, at Cycle 3 Day 1 (each cycle is 21 days) and at the end of treatment for 2 years
  Microbiome analysis on stool samples will be assessed through whole metagenomics sequencing in order to evaluate roles of microbiome communities in immunotherapy.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre Henri Becquerel, Rouen
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse